CLINICAL TRIAL: NCT03583827
Title: Motor Learning of Stroke Patients in Virtual Environments: Randomized Controlled Clinical Trial
Brief Title: Motor Learning of Stroke Patients in Virtual Environments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Rio Grande do Norte (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Tania Campos, Associate Professor and Researcher, Universidade Federal do Rio Grande do Norte
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 475182/2012-0
Record Dates: First submitted 2018-06-07; First posted 2018-07-11 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Stroke; Stroke Sequelae
Keywords: Cerebrovascular disorders; Upper extremity; Paresis; Electroencephalography; Psychomotor Performance
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders; Paresis

STUDY DESIGN:
Intervention Model Description: Eighty unilaterally brain injured right-handed patients, with lesion time of 6 months or more, aged 70 years or younger, 40 with left-brain and 40 with right-brain injury, will take part in the study. They will be randomly divided into a control group (GC), which will undergo conventional therapy and an experimental group (EG), which will be submitted to conventional and virtual reality training using the game virtual. The study will also include 40 healthy individuals matched for age, sex, schooling and hand laterality.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): Experimental group patients will be submitted to conventional therapy for 30 minutes and training of the affected upper limb using virtual reality, which will last 20 minutes over twelve sessions (4 weeks).
  Interventions: Other: Virtual reality; Other: Conventional physical therapy
- Control Group (Active Comparator): The control group will undergo 30 minutes of Conventional physical therapy in twelve sessions (4 weeks).
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Other: Virtual reality — Virtual reality is a simulation of the real world generated by computer software and experienced by users via a man-machine interface, providing them with intensive repetition of complex tasks, directed by visual and auditory stimuli, creating dynamic individual-task interaction, a motivating environment and immediate feedback on performance and results, stimulating motor skill learning and motor control of complex behaviors.
  Other Names: Virtual game
  Arms: Experimental Group
Other: Conventional physical therapy — Exercises of stretching and strengthening of the upper and lower limbs, as well as coordination, gait and balance.
  Other Names: Traditional physical therapy

SUMMARY:
The aim of this study is to assess the motor learning of patients with chronic stroke in virtual environments. Half the patients will undergo conventional therapy and half virtual reality training using virtual game. The study will also include healthy individuals matched for age, sex, schooling and hand laterality.

DETAILED DESCRIPTION:
Stroke is the main cause of long-term disability in adults and motor learning is vital for recovering from motor sequelae. A number of approaches have been proposed to promote motor learning, including virtual reality, which simulates a real world environment and is based on the assumption that skills acquired in a virtual world will be transferred to the real world. Virtual reality induces use-dependent plastic changes in response to stimulation of higher motor areas, recruiting the memory system containing stored motor programs. As such, these interactive interventions of virtual reality are based on the idea that stimulating the action processing system activates the cortical areas involved in movement execution.

These game characteristics allow activation of the mirror neuron system during the execution or observation of actions. Recent evidence suggests an important role for this neuron system in the improvement or motor recovery of patients. In this respect, observing an action in association with physical training may enhance the effects of motor training on the recovery of patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with the first episode of stroke, confirmed by medical imaging examination, unilateral brain injury, lesion time of at least 6 months;
* Right-handed and able to complete the assessment instruments;
* Individuals with affected upper limb movement skills, such as drinking water from a glass;
* Subjects able to remain in the orthostatic position, with or without gait assistive device.

Exclusion Criteria:

* Unilateral neglect and uncorrected primary auditory or visual impairment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-02-10 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Change the angle of movement | Change from baseline until 30 days.
  Angle of extension of the elbow joint (in degrees) measured before and after the intervention.

SECONDARY OUTCOMES:
Change the EEG power of alpha and beta waves | Change from baseline until 30 days.
  EEG power of alpha and beta waves (uV2) measured before and after the intervention.
Change the Absolute error | Change from 15 trials during 20 minutes over twelve sessions (4 weeks).
  Absolute error evaluated by score which may vary from 0 (no error, the dart hits the central target) to 5 (maximum error, the dart does not hits the target).

CONTACTS AND LOCATIONS:
Overall Officials: Tania F Campos, PhD, Study Director — Universidade Federal do Rio Grande do Norte
Locations (1):
- Department of Physical Therapy-Federal University of Rio Grande do Norte, Natal, Rio Grande do Norte, Brazil

IPD SHARING:
Plan to Share IPD: No